CLINICAL TRIAL: NCT00159406
Title: Laser Prostatectomy for Benign Prostatic Hyperplasia: A Registry and Database
Brief Title: Laser Prostatectomy Database and Registry
Status: Active, not recruiting | Type: Observational
Sponsor: Indiana Kidney Stone Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 03-095
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Benign Prostatic Hyperplasia; Enlarged Prostate
Keywords: BPH treatment; Laser Prostatectomy; Treatment of enlarged Prostates; BPH
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Registries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cohort: Registry and Database
  Interventions: Other: Registry and Database

INTERVENTIONS:
Other: Registry and Database — Data Collection

SUMMARY:
STATEMENT OF PURPOSE:

Transurethral resection of the prostate (TURP) is the standard surgical intervention for obstructive benign prostatic hyperplasia (BPH) in all but the largest of glands, which are typically treated with open simple prostatectomy. Recently, new generation lasers (holmium and potassium titanyl phosphate [KTP]) have been utilized for BPH treatment. Long-term follow-up of laser prostatectomy outcomes must be documented to fully characterize the degree of voiding improvement achievable by these new techniques, the durability of these outcomes, and the safety profiles of these procedures.

DETAILED DESCRIPTION:
Benign prostatic hyperplasia (BPH) affects over 40% of men over the age of 60 (Kirby RS, 2000). For patients with significant obstructive symptoms which are not helped by medical therapy, surgical intervention is instituted. Transurethral resection of the prostate (TURP), an endoscopic procedure where prostate tissue is sequentially removed with an electrocautery loop, remains the gold standard to which other surgical therapies are compared. Unfortunately, TURP is associated with significant patient morbidity such as blood loss and dilutional hyponatremia, especially when resection times are prolonged (Mebust WK et al, 1989).

Because of the long resection times and increased morbidity risks involved in patients with extremely large prostate glands, open simple prostatectomy was traditionally employed in place of TURP to remove the obstructing adenoma tissue. However, the patient could still expect a prolonged hospital stay and a high likelihood of post-operative transfusion.

Many alternative surgical treatments for BPH have been developed in an attempt to minimize the morbidity profile of the more traditional surgical approaches. New generation holmium (2140 nm wavelength) and KTP (532 nm wavelength) lasers now offer a minimally invasive alternative to BPH treatment broadly termed laser prostatectomy. Within the category of laser prostatectomy, two distinctly separate techniques have been developed. The first, laser ablation, involves the vaporization of obstructive prostate tissue. Effective ablation can be achieved with either the holmium or KTP laser. Previous groups have reported favorable outcomes with minimal associated morbidity when treating smaller prostates with the laser ablation technique (Hai MA and Malek RS, 2003).

The properties of the holmium laser also enable it to cut soft tissue while maintaining hemostasis, such that it can be utilized for dissecting entire prostatic lobes away from the prostatic capsule. This procedure has been termed holmium laser enucleation of the prostate (HoLEP), and it can be performed on even the largest of glands to duplicate the results of open simple prostatectomy with much less morbidity (Gilling PJ et al, 2000 and Moody JA and Lingeman JE, 2001).

We have performed both holmium and KTP prostate ablations and have had extensive clinical experience with the HoLEP procedure. Our impressions of the various laser prostatectomy procedure outcomes appear to substantiate the findings of the aforementioned studies. However, extended follow-up of patients undergoing laser prostatectomies and documentation of their outcomes and associated complications must be done in order to support the initial conclusions of the previous investigators.

SPECIFIC AIMS:

To review the outcomes of our population of patients with BPH who have undergone laser prostatectomy. We hypothesize that the long-term improvements in voiding parameters achieved by these new laser procedures will compare favorably and perhaps be better than results previously reported for TURP or, in the case of larger glands, open simple prostatectomy. In addition, the adverse events/complication profile of the laser procedures should be better than those of the traditional treatments. Once all retrospective data has been reviewed, we will continue to collect outcome data on a prospective basis.

ELIGIBILITY:
Inclusion Criteria:

* Patients of IU Health Physicians Urology in Indianapolis, Indiana
* Male patients over the age of 18 with benign prostatic hyperplasia requiring surgical intervention for symptomatic relief.

Exclusion Criteria:

* Patients unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of IU Health Physicians Urology who are already scheduled to undergo a laser prostatectomy
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2003-10; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Time to achieve continence | Ongoing

SECONDARY OUTCOMES:
No urinary retention | ongoing
AUA SS | ongoing
Bother index score | ongoing
Decreased PSA | ongoing
Decreased prostate size | ongoing
Minimal complications | ongoing

CONTACTS AND LOCATIONS:
Overall Officials: James E Lingeman, MD, Principal Investigator — IU Health Physicians Urology
Locations (1):
- IU Health Methodist Hospital, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Tinmouth WW, Habib E, Kim SC, Kuo RL, Paterson RF, Terry CL, Elhilali M, Lingeman JE. Change in serum prostate specific antigen concentration after holmium laser enucleation of the prostate: a marker for completeness of adenoma resection? J Endourol. 2005 Jun;19(5):550-4. doi: 10.1089/end.2005.19.550. PMID 15989443
- [Result] Kuo RL, Paterson RF, Kim SC, Siqueira TM Jr, Elhilali MM, Lingeman JE. Holmium Laser Enucleation of the Prostate (HoLEP): A Technical Update. World J Surg Oncol. 2003 Jun 6;1(1):6. doi: 10.1186/1477-7819-1-6. PMID 12818001
- [Result] Kuo RL, Kim SC, Lingeman JE, Paterson RF, Watkins SL, Simmons GR, Steele RE. Holmium laser enucleation of prostate (HoLEP): the Methodist Hospital experience with greater than 75 gram enucleations. J Urol. 2003 Jul;170(1):149-52. doi: 10.1097/01.ju.0000070686.56806.a1. PMID 12796668
- [Result] Peterson MD, Matlaga BR, Kim SC, Kuo RL, Soergel TM, Watkins SL, Lingeman JE. Holmium laser enucleation of the prostate for men with urinary retention. J Urol. 2005 Sep;174(3):998-1001; discussion 1001. doi: 10.1097/01.ju.0000170230.26743.e4. PMID 16094022
- [Result] Kim SC, Matlaga BR, Kuo RL, Watkins SL, Kennett KM, Gilling PJ, Lingeman JE. Holmium laser enucleation of the prostate: a comparison of efficiency measures at two institutions. J Endourol. 2005 Jun;19(5):555-8. doi: 10.1089/end.2005.19.555. PMID 15989444
- [Result] Kuo RL, Paterson RF, Siqueira TM Jr, Watkins SL, Simmons GR, Steele RE, Lingeman JE. Holmium laser enucleation of the prostate: morbidity in a series of 206 patients. Urology. 2003 Jul;62(1):59-63. doi: 10.1016/s0090-4295(03)00124-9. PMID 12837423